CLINICAL TRIAL: NCT06220331
Title: Intensity Lenses Post Operation Standard of Care Visits - Data Collection.
Brief Title: Data Collection After Intensity IOL Implantations
Status: Completed | Type: Observational
Sponsor: Hanita Lenses (Industry)
Responsible Party: Sponsor
Other Study IDs: RT-IN1
Record Dates: First submitted 2024-01-14; First posted 2024-01-23 (Actual); Last update posted 2024-01-23 (Actual); Status verified 2024-01

CONDITIONS: Cataract
Keywords: Intra Ocular Lens; Intensity SL; Hanita Lenses; Cataract
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Elder patients diagnosed with cataract: Patients that diagnosed with cataract and had implantation with Hanita Intensity IOL or Intensity Toric Lenses in the clinic participating in the study.
  Interventions: Device: Intra Ocular Lens

INTERVENTIONS:
Device: Intra Ocular Lens — Intensity SL Intra Ocular Lens

SUMMARY:
Hanita Lenses new Intensity IOL and Intensity Toric were been designed to have very high efficiency of light leading to a high MTF, wide focal ranges of far, intermediate and near vision and minimal loss of light energy. The main purpose of this study is to collect existing post-operative data based on standard of care follow up visits at the clinic.

DETAILED DESCRIPTION:
Different multifocal intraocular lens (MIOL) designs have been used for more than 25 years1. Unlike conventional mono focal intraocular lenses (IOLs), which bend light to a single focus point on the retina, MIOLs are designed to help patients to see at varying distances using different points of focus2. MIOLs used in clinical practice were either refractive initially, or later diffractive in their optical design. Refractive MIOLs incorporate a lens optic with different optical powers in different parts of the lens, while diffractive MIOLs use diffractive steps on the lens to distribute light rays into two or more principal foci. Irrespective of the design type, however, all MIOLs involve some form of optical compromise and a process of neuroadaptation for the patient.

Intensity SL intraocular lenses (IOLs) represent the latest in premium lens technology. Intensity SL lenses provide clear vision at all distances - from near to far - thus offering the best chance of true spectacle independence.

Despite the promising results obtained with the latest generation of MIOLs, many surgeons remain reluctant to implant these lenses. Visual symptoms such as glare and haloes, reduced contrast sensitivity and night vision problems are all known complications of multifocal implants and have served to hamper wider acceptance of these IOLs4.

Hanita Lenses new Intensity IOL and Intensity Toric were been designed to have very high efficiency of light leading to a high MTF, wide focal ranges of far, intermediate and near vision and minimal loss of light energy. The main purpose of this study is to collect existing post-operative data based on standard of care follow up visits at the clinic.

ELIGIBILITY:
Inclusion Criteria:

* Patient over the age of 18
* Patient who underwent bilateral implantations with Hanita Lenses Intensity IOL

Exclusion Criteria:

* Patients who don't have any follow up visits after implantation

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Men and women that had implantation with Hanita Intensity IOL or Intensity Toric Lenses in the clinic participating in the study. The patients that suffered from cataract and operated with implantation of Hanita Intensity MIOL or Intensity Toric MIOL in the clinic participating in the study.
Sampling Method: Non-Probability Sample
Enrollment: 31 (Actual)
Dates: Start 2023-07-13 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
The aim of this study is to evaluate performance of Hanita Lenses Intensity SL IOL. | 1-3 months
  Performance of the IOL will be evaluated by assessing the defocus Curve and visual acuity for far, intermediate and near distance after Intensity SL IOL implantation.

SECONDARY OUTCOMES:
The second aim of this study is to evaluate the visual phenomena post-operation. | 1-3 months
  Visual phenomena will be evaluated by asking the patients about halos ang glares

CONTACTS AND LOCATIONS:
Locations (1):
- Consejo Argentino de Oftalmología, Buenos Aires, Argentina

IPD SHARING:
Plan to Share IPD: No